CLINICAL TRIAL: NCT00391794
Title: Efficacy of Early Stage Alzheimer's Support Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rebecca Logsdon, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29920-J; 5R01AG023091 (NIH); 06-1324-G01 (Other: UW Human Subjects Division); 5R01AG023091-02 (NIH); 1A0131
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Memory Loss; Alzheimer's Disease; Dementia
Keywords: Memory; Alzheimer's disease; Dementia; Support Group; Psychosocial
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESSG (Experimental): eight weekly 90-minute sessions
  Interventions: Behavioral: Early Stage Memory Loss Support Group
- ES (Active Comparator): one 4-hour educational program
  Interventions: Behavioral: Educational Seminar

INTERVENTIONS:
Behavioral: Early Stage Memory Loss Support Group — 8 week support group led by trained facilitators
  Other Names: ESSG
  Arms: ESSG
Behavioral: Educational Seminar — 4 hour education session led by trained facilitators
  Other Names: ES
  Arms: ES

SUMMARY:
The purpose of this study is to evaluate the impact of an Early Stage Memory Loss Support Group (ESSG) and Education Seminar (ES) on quality of life, mood, social support, distress about memory loss, and interpersonal relationships of memory loss participants and their caregivers.

DETAILED DESCRIPTION:
With recent advances in diagnostic procedures and treatment options, many individuals with AD are now diagnosed early in the disease. Early diagnosis has many benefits: treatment can be started sooner, legal and financial planning can be addressed while the individual is able to participate in decision-making, and support services can be mobilized earlier. However, early diagnosis may also have negative consequences for the diagnosed individual's quality of life. Thus, diagnosis creates an obligation to help individuals and their families learn more about AD and cope with the impact of the diagnosis. Many Alzheimer's Association chapters have begun providing early stage support groups that focus on enhancing quality of life for participants and their caregivers. Anecdotal reports suggest that these groups improve quality of life of participants, but some individuals may also experience decreases in quality of life associated with stress, depression, or family conflict as a result of discussing current and future losses in the group. Thus, there is a need to systematically evaluate the benefits of these groups.

This study will evaluate and compare the efficacy of a structured, 8-session Early Stage Support Group intervention (ESSG) and a half-day Education Seminar (ES). Participants with early stage memory loss and their caregivers will be randomly assigned to either ESSG or ES. Both are presented by the Alzheimer's Association Western & Central Washington State Chapter.

ELIGIBILITY:
Inclusion Criteria:

* Dementia diagnosis confirmed by primary care physician
* Early stage dementia, defined as a Mini Mental State Exam score of 18 or higher, and a Clinical Dementia Rating of 1 or less
* Care partner who will attend groups and complete study assessments
* Aware of memory loss (verbally acknowledges memory loss and/or expresses concern about memory)
* Comfortable in a group separate from family members
* No significant history of mental illness (no hospitalization or medication for psychotic disorder within the past 2 years)
* Consent to research participation (participant, care partner, legal representative)
* Remain in the community for the 6 month duration of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Quality of life | baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
Mood | baseline, 3 months, and 6 months
Social support | baseline, 3 months, and 6 months
Family Relationships | baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Logsdon, PhD., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Goldsilver PM, Gruneir MR. Early stage dementia group: an innovative model of support for individuals in the early stages of dementia. Am J Alzheimers Dis Other Demen. 2001 Mar-Apr;16(2):109-14. doi: 10.1177/153331750101600206. PMID 11302071
- [Background] Quayhagen MP, Quayhagen M, Corbeil RR, Hendrix RC, Jackson JE, Snyder L, Bower D. Coping with dementia: evaluation of four nonpharmacologic interventions. Int Psychogeriatr. 2000 Jun;12(2):249-65. doi: 10.1017/s1041610200006360. PMID 10937544
- [Background] Snyder L, Quayhagen MP, Shepherd S, Bower D. Supportive seminar groups: an intervention for early stage dementia patients. Gerontologist. 1995 Oct;35(5):691-5. doi: 10.1093/geront/35.5.691. PMID 8543229
- [Background] Zarit SH, Femia EE, Watson J, Rice-Oeschger L, Kakos B. Memory Club: a group intervention for people with early-stage dementia and their care partners. Gerontologist. 2004 Apr;44(2):262-9. doi: 10.1093/geront/44.2.262. PMID 15075423